CLINICAL TRIAL: NCT01903408
Title: Prostate and Whole Pelvis Irradiation With Integrated-boost Intensity-modulated Radiotherapy (IMRT) After Neoadjuvant Antihormonal Treatment - a Phase II Trial
Brief Title: Radiotherapy of the Prostate and the Pelvic Lymph Nodes After Neoadjuvant Antihormonal Treatment
Acronym: PLATIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Klaus Tschira Stiftung gGmbH (Unknown)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Principal Investigator, Heidelberg University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Klaus Tschira 00.153.2009; ARO 2009-05 (Registry Identifier: ARO)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1: Boost to prostate (Other): IMRT of the pelvic lymphatic drainage (51 Gy) and integrated boost to the prostate (76.5 Gy) in 34 fractions Arm finished recruitment and follow-up
  Interventions: Radiation: Intensity-modulated radiotherapy of the pelvic lymph nodes using SIB
- Arm 2: Boost to prostate and lymph node metastases (Other): IMRT of the pelvic lymphatic drainage (51 Gy), SIB to the prostate (76.5 Gy) & pelvic lymph node mets (61.2 Gy) in 34 Fx
  Interventions: Radiation: Intensity-modulated radiotherapy of the pelvic lymph nodes using SIB
- Arm 3: Boost to prostate bed (Other): IMRT of the pelvic lymphatic drainage (51 Gy) and integrated boost to the prostate bed (68 Gy) in 34 fractions Arm finished recruitment and follow-up and is published
  Interventions: Radiation: Intensity-modulated radiotherapy of the pelvic lymph nodes using SIB
- Arm 4: Boost to prostate bed and lymph node metastases (Other): IMRT of the pelvic lymphatic drainage (51 Gy), SIB to the prostate bed 68 Gy) & lymph node metastases (61.2 Gy) in 34 Fx
  Interventions: Radiation: Intensity-modulated radiotherapy of the pelvic lymph nodes using SIB
- Arm 5: Boost to lymph node metastases (Other): Patients with previous irradiation of the prostate bed: IMRT of the pelvic lymphatic drainage (46.8 Gy) above the previous treatment fields, SIB to lymph node metastases (63.2 Gy) in 26 Fx
  Interventions: Radiation: Intensity-modulated radiotherapy of the pelvic lymph nodes using SIB

INTERVENTIONS:
Radiation: Intensity-modulated radiotherapy of the pelvic lymph nodes using SIB — The intervention is the use of modern radiation techniques with simultaneous integrated boost (SIB)

SUMMARY:
For patients with prostate cancer and a high risk of lymph node involvement or confirmed pelvic lymph node metastases, radiotherapy of the whole pelvis is a treatment option. However, conventional radiotherapy of the pelvis has limited by gastrointestinal and urogenital side effects. The PLATIN trial investigates an intensity-modulated radiotherapy of the pelvic lymphatic drainage that spares small bowel, bladder and rectum. A higher dose is given during each session to the prostate or the prostate bed and to confirmed lymph node metastases. Prior to radiotherapy, two months of neoadjuvant antihormonal treatment are required, and continuation during radiotherapy and for a further two years are strongly recommended.

DETAILED DESCRIPTION:
The PLATIN trial is designed as a prospective, non-randomized, five-arm trial. Arm 1: Definitive radiotherapy of the pelvic lymphatic drainage with integrated boost to the prostate.

Arm 2: As arm 1, with additional boost to macroscopic lymph node metastases. Arm 3: Postoperative radiotherapy of the pelvic lymphatic drainage with integrated boost to the prostate bed.

Arm 4: As arm 3, additional boost to macroscopic lymph node metastases. Arm 5: Patients with previous radiotherapy to the prostate bed. Radiotherapy of the pelvic lymphatic drainage above the previous treatment fields with integrated boost to macroscopic lymph node metastases.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed prostate cancer with Gleason Score
* risk of lymph node involvement >20% (according to Roach Formula), pelvic lymph node metastases in CT/MRI or histologically confirmed lymph node involvement
* Karnofsky Index >/= 70%
* age 18-75 years
* neoadjuvant antihormonal treatment for 2 months, continuation until the end of radiotherapy
* written informed consent

Exclusion Criteria:

* stage IV (distant metastases)
* lymph node metastases outside the pelvis
* rising prostate-specific antigen (PSA) under antihormonal treatment
* severe wound complications after laparatomy
* severe lymph edema of the legs, elephantiasis, postthrombotic syndrome
* decompensated comorbidity of the lungs, heart, metabolic system, hematopoetic system or kidneys, coagulopathy
* history of other malignancy within the last 5 years (except for basal cell carcinoma or squamous carcinoma of the skin)
* previous irradiation of the pelvic lymph nodes
* concurrent participation in a clinical trial that might influence the results of either trial

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Rate of safe feasibility (SDR) | 2 years
  Proportion of treatments begun as planned without grade 3-4 NCI common toxicity criteria adverse events (CTC AE) or treatment disruption among all patients that fulfill inclusion criteria and have been treated according to trial protocol for at least a week.

SECONDARY OUTCOMES:
Biochemical recurrence free survival | 2 years
Quality of Life | 2 years
  Measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, Prof. Dr., Principal Investigator — University Hospital Heidelberg, Department of Radiation Oncology
Locations (1):
- Department of Radiation Oncology, University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Result] Habl G, Katayama S, Uhl M, Kessel KA, Edler L, Debus J, Herfarth K, Sterzing F. Helical intensity-modulated radiotherapy of the pelvic lymph nodes with a simultaneous integrated boost to the prostate--first results of the PLATIN 1 trial. BMC Cancer. 2015 Nov 7;15:868. doi: 10.1186/s12885-015-1886-5. PMID 26547188
- [Result] Katayama S, Habl G, Kessel K, Edler L, Debus J, Herfarth K, Sterzing F. Helical intensity-modulated radiotherapy of the pelvic lymph nodes with integrated boost to the prostate bed - initial results of the PLATIN 3 Trial. BMC Cancer. 2014 Jan 14;14:20. doi: 10.1186/1471-2407-14-20. PMID 24422782
- [Result] Koerber SA, Winter E, Katayama S, Slynko A, Haefner MF, Uhl M, Sterzing F, Habl G, Schubert K, Debus J, Herfarth K. Elective Node Irradiation With Integrated Boost to the Prostate Using Helical IMRT-Clinical Outcome of the Prospective PLATIN-1 Trial. Front Oncol. 2019 Aug 13;9:751. doi: 10.3389/fonc.2019.00751. eCollection 2019. PMID 31456941